CLINICAL TRIAL: NCT04603300
Title: Oral Mucosal Escalation Goal Assessment (OMEGA) Study: A Randomized Placebo-Controlled Phase 1 Study of the Safety and Feasibility of Up-titration With INT301 in Adults With Sensitivity to Peanut
Brief Title: OMEGA Study: A Study of the Safety and Feasibility of Up-titration With INT301 in Adults With Sensitivity to Peanut
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intrommune Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INT301-101
Record Dates: First submitted 2020-09-25; First posted 2020-10-26 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Peanut Allergy
Keywords: Peanut allergy; Food allergy; Desensitization; Allergy Immunotherapy; OMIT; OIT; EPIT; SLIT; Oral Mucosal Immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind is controlled by IWRS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active treatment (Active Comparator): INT301 dosing as determined by cohort assignment
  Interventions: Drug: INT301
- Placebo (Placebo Comparator): Placebo as determined by cohort assignment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INT301 — INT301 is an allergy immunotherapy delivered in the form of a fully functional toothpaste
  Arms: Active treatment
Drug: Placebo — Fully functional toothpaste containing no immunotherapy agents
  Arms: Placebo

SUMMARY:
This is a phase 1, multi-center, randomized, double-blind, placebo-controlled study in adult participants with peanut allergy. Participants will be randomized in a 3:1 ratio to receive either an escalating dose of INT301 or placebo. The treatment group will be blinded to the investigator, participants, and the Intrommune study team.

ELIGIBILITY:
Inclusion Criteria:

Participant must be 18-55 years of age inclusive, at the time of signing the informed consent.

Female participants of childbearing potential or male participants with female partners of child-bearing potential must utilize highly effective birth control method(s) throughout the study and for 30 days after the final dose of study drug. Acceptable methods of contraception include: complete abstinence, male or female condoms with spermicide, oral or implanted contraceptives, or vasectomy.

For female participants of child-bearing potential: Negative serum beta human chorionic gonadotrophin (HCG) pregnancy test at screening.

Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Meets at least one of the following conditions

* Positive skin prick test (SPT) (wheal at least 3 mm greater than control) AND/OR Peanut specific IgE >0.35 kU/L
* Convincing clinical history of allergic reaction to peanut within 1 hour of ingestion for at least 3 months prior to screening.
* Failed an oral food challenge (OFC) of < 100mg of peanut protein at screening.
* Participant willing and able to undergo the procedures required by the protocol, including, assessment completion, protocol compliance, and participation in the placebo dosing period(s).

Exclusion Criteria:

* History of severe anaphylaxis to peanut, defined as hypoxia, hypotension, or neurologic compromise (cyanosis or oxygen saturations < 92% at any stage, hypotension, confusion, collapse, loss of consciousness, or incontinence)
* Significant medical condition (e.g., liver, kidney, gastrointestinal, cardiovascular, hematologic, or pulmonary disease) which would make the subject unsuitable for induction of food reactions
* Eosinophilic or other inflammatory (e.g. celiac) gastrointestinal disease
* Psychiatric disorders that the Investigator believes will interfere with study assessments
* Uncontrolled asthma, defined by at least one of the following conditions:

  * - FEV1 <80% of predicted, or ratio of FEV1 to forced vital capacity (FEV1/FVC) <75% of predicted, with or without controller medications.
  * - Inhaled corticosteroids (ICS) dosing of >500mcg daily fluticasone (or equivalent ICS based on NHLBI dosing chart.
  * - One hospitalization in the past year for asthma
  * - An ER visit for asthma within six months prior to screening
* Planned dental surgery during from screening until study exit
* Moderate or advanced periodontal disease.
* Current pregnancy or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of INT301 compared to placebo in adult peanut allergic participants as measured by dose escalation during study. | Forty-eight weeks
  Percentage of participants able to consistently tolerate the protocol-specified highest dose; Incidence of systemic and non-systemic adverse reactions.

SECONDARY OUTCOMES:
To evaluate pharmacologic requirements as interventions for peanut allergic participants experiencing adverse events on INT301. | Forty-eight weeks
  Number of participants requiring treatment for systemic reactions related to experimental treatment or placebo; Number of adverse events requiring treatment for systemic reactions related to experimental treatment or placebo; Adherence to study treatment.
To determine the maximally tolerated dose during the up-dosing phase for adults. | Twenty-six weeks
  Dose amount tolerated without AEs requiring discontinuation for each participant.

OTHER OUTCOMES:
To explore changes in peanut-specific IgG4, IgA, and IgE levels in participants (exploratory outcome). | Forty-eight weeks
  Change from baseline of peanut-specific IgG4, IgA, and IgE in study subjects (exploratory outcome)
To explore changes in patient response to oral food challenge pre-treatment and post treatment. | Forty-eight weeks
  Change from baseline of tolerated amount of peanut protein

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hudson-Essex Allergy, Belleville, New Jersey
  - Weiss Medical, Riverdale, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger WE, Faris N, Weinstein M, Wilding GE, Berglund E. Randomized, placebo-controlled, phase 1 safety study of oral mucosal immunotherapy in adults with peanut allergy. Ann Allergy Asthma Immunol. 2025 Apr;134(4):448-456. doi: 10.1016/j.anai.2025.01.013. Epub 2025 Jan 20. PMID 39842774